CLINICAL TRIAL: NCT06146062
Title: Effects of Intravascular Administration of Mesenchymal Stromal Cells Derived from Wharton's Jelly of the Umbilical Cord on Systemic Immunomodulation and Neuroinflammation After Traumatic Brain Injury.
Acronym: TRAUMACELL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211509; 2021-006873-50 (EudraCT Number)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: use of placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Final product is a MSC solution at the concentration of 2.10^6/kg in 150 mL of NaCl 0.9% and human albumin 0.5%, conditioned aseptically and identified for IV administration.
  3 injections one week apart.
  Interventions: Drug: Mesenchymal Stromal Cells (MSC)
- control (Placebo Comparator): The placebo will be a solution of NaCl 0.9% 3 injections one week apart.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mesenchymal Stromal Cells (MSC) — 3 injections one week apart
  Arms: Intervention
Drug: placebo — 3 injections one week apart
  Arms: control

SUMMARY:
Traumatic brain injuries (TBI) are one of the leading causes of death and disability worldwide. These patients are burdened by physical, cognitive, and psychosocial deficits, leading to an important economic impact for society. Treatments for TBI patients are limited and none has been shown to provide prolonged and long-term neuroprotective or neurorestorative effects. TBI related disability is linked to the severity of the initial injury but also to the following neuroinflammatory response which may persist long after the initial injury.

Moreover, a growing body of evidence suggests a link between TBI-induced neuro-inflammation and neurodegenerative post traumatic disorders. Consequently, new therapies triggering immunomodulation and promoting neurological recovery are the subject of major research efforts.

In this context, mesenchymal cell-based therapies are currently investigated to treat various neurological disorders due to their ability to modulate neuroinflammation and to promote simultaneous neurogenesis, angiogenesis, and neuroprotection.

Clinical trials using intravenous MSC have been conducted for various pathologies, all these studies showing a good safety profile.

The hypothesis of the study is that intravenous repeated treatment with MSC derived from Wharton's Jelly of the umbilical cord may be associated with a significant decrease of post-TBI neuroinflammation and improvement of neuroclinical status.

The main objective of the study is to evaluate the effect of iterative IV injections of MSC on post-traumatic neuroinflammation measured in corpus callosum by PET-MRI at 6 months in severe brain injured patients unresponsive to simple verbal commands 5 days after sedation discontinuation.

DETAILED DESCRIPTION:
Traumatic brain injuries (TBI) are one of the leading causes of death and disability worldwide. These patients are burdened by physical, cognitive, and psychosocial deficits, leading to an important economic impact for society. Treatments for TBI patients are limited and none has been shown to provide prolonged and long-term neuroprotective or neurorestorative effects. TBI related disability is linked to the severity of the initial injury but also to the following neuroinflammatory response which may persist long after the initial injury.

Moreover, a growing body of evidence suggests a link between TBI-induced neuro-inflammation and neurodegenerative post traumatic disorders. Consequently, new therapies triggering immunomodulation and promoting neurological recovery are the subject of major research efforts.

In this context, mesenchymal cell-based therapies are currently investigated to treat various neurological disorders due to their ability to modulate neuroinflammation and to promote simultaneous neurogenesis, angiogenesis, and neuroprotection. Indeed, several experimental studies have reported that human umbilical cord-derived mesenchymal stromal cells (MSC) have the ability to improve neurological outcomes and recovery in cerebral injury animal models, including TBI.

Clinical trials using intravenous MSC have been conducted for various pathologies, all these studies showing a good safety profile. In TBI, small clinical trials using different modalities for administration of mesenchymal cells are available but none about MSC derived from Wharton's Jelly of the umbilical cord.

The hypothesis of the study is that intravenous repeated treatment with MSC derived from Wharton's Jelly of the umbilical cord may be associated with a significant decrease of post-TBI neuroinflammation and improvement of neuroclinical status.

The main objective of the study is to evaluate the effect of iterative IV injections of MSC on post-traumatic neuroinflammation measured in corpus callosum by PET-MRI at 6 months in severe brain injured patients unresponsive to simple verbal commands 5 days after sedation discontinuation.

ELIGIBILITY:
20 healthy volunteers will be included for MRI normalization Volunteer eligibility criteria

Inclusion criteria :

* Age 18-50 years
* ASA 1 classification (healthy patient)

Exclusion criteria :

* Lack of written consent
* Neurological history likely to alter the image (epilepsy, transient ischaemic attack, meningitis, head trauma)
* Vulnerable person according to article L1121-6 of the CSP
* Protected adult person
* No affiliation to a social security regime
* Pregnancy
* Contraindication for MRI and PET-MRI

  * patients with Pacemaker and defibrillator
  * MR-incompatible prosthetic heart valve
  * Metallic intraocular, intra cerebral or intra medullary foreign bodies
  * Implantable neurostimulation systems
  * Cochlear implants/ear implant
  * Metallic fragments such as bullets, shotgun pellets, and metal shrapnel
  * Cerebral artery aneurysm clips
  * Ventriculo peritoneal shunt with metallic component generating significant artefacts on the MR sequence
  * Catheters with metallic components (Swan-Ganz catheter)
  * Patient unable to remain supine and motionless during the duration of the examination

    68 severe TBI patients with the following inclusion and exclusion criteria will be included"

Patient Inclusion criteria

* Age 18-50 years
* Severe TBI defined by:

  * Glasgow score <12 within the 48 first hours,
  * Brain traumatic lesion on CT scan,
  * Need for intracranial pressure monitoring
* No other significant organ trauma (AIS <2)
* Unresponsive to verbal commands 5 days after sedation discontinuation, for whom, after usual clinical and paraclinical evaluation there has been no decision to interrupt active therapies within 10 days after sedation discontinuation
* Written consent signed by the close relative

Patient Exclusion criteria

* History of disease or treatment impairing current or previous year immunity function ( hematologic disease (leukemia, myeloma), viral disease affecting immunity (like HIV), immunological treatment (corticoid, anti rejection medication, anti TNFα, chemotherapy)
* History of severe neurological or psychiatric disease likely to alter neurological assessment
* HTAP > grade III OMS/WHO
* Ongoing uncontrolled infection with organ failure (septic shock, ARDS) including those due to severe COVID-19
* Platelets <100 G/L or <100000/μL, Hb <8 g/dL, lymphocytes count <1.5 G/L or 1500 μL , neutrophils count < 2.5G/L or <2500/μL, , creatinin > 100 μmol/L
* Liver function abnormalities (bilirubin> 2.5mg / dL or transaminases> 5x the ULN). Patients with Gilbert's disease are eligible if liver tests are normal excluding bilirubinemia
* Known HIV seropositivity
* Neoplasia ongoing or treated in the 3 years before screening
* Bone marrow transplant recipient
* History of transfusion reaction or hypersensitivity
* Pregnancy
* Contraindication for MRI and PET-MRI:

  * Patient with Pacemaker and defibrillator
  * MR-incompatible prosthetic heart valve o Metallic intraocular, intra cerebral or intra medullary foreign bodies
  * Implantable neurostimulation systems o Cochlear implants/ ear implant
  * Metallic fragments such as bullets, shotgun pellets, and metal shrapnel
  * Cerebral artery aneurysm clips
  * Ventriculo peritoneal shunt with metallic component generating significant artefacts on the MR sequence
  * Catheters with metallic components (Swan-Ganz catheter)
  * Patient unable to remain supine and motionless during the duration of the examination
* Participation in another interventional clinical trial of an investigational therapy within 30 days of consent
* No affiliation to a social security regime
* Vulnerable person according to article L1121-6 of the CSP
* Protected adult person

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
effect of iterative IV injections of WJ-UC-MSC on post-traumatic neuroinflammation | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in corpus callosum (Region of Interest, ROI) measured by dynamic PET-MRI

SECONDARY OUTCOMES:
radiological markers from PET-MRI_1 | 6 months after the last injection
  The regional fractional anisotropy (FA) from DTI acquisition of PET-MRI
radiological markers from PET-MRI_2 | 6 months after the last injection
  The mean diffusibility (MD) from DTI acquisition of PET-MRI
Treatment feasibility | at the third injection
  number of treatments administrated to the patient
Neurological clinical Score M6 | 6 months after the last injection
  Glasgow Outcome Scale-Extended
Neurological clinical Score M12 | 12 months after the last injection
  Glasgow Outcome Scale-Extended
cognitive assessment M6 | 6 months after the last injection
  MOCA scale
cognitive assessment M12 | 12 months after the last injection
  MOCA scale
short term Tolerance D10 | 10 days after the last injection
  Common Terminology Criteria for Adverse Events
long term Tolerance M6 | 6 months after the last injection
  Common Terminology Criteria for Adverse Events
long term Tolerance M12 | 6 months after the last injection
  Common Terminology Criteria for Adverse Events
neuroinflammation of pericontusional | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in pericontusional
neuroinflammation of grey matter | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in grey matter
neuroinflammation of white matter | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in white matter
neuroinflammation of frontal area | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in frontal area
neuroinflammation of parietal area | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in parietal area
neuroinflammation of occipital area | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in occipital area
neuroinflammation of hippocampus | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in hippocampus,
neuroinflammation of thalamus | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in thalamus,
neuroinflammation of mesencephalus | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in mesencephalus
neuroinflammation of cerebellum | 6 months after the last injection
  [18F]-DPA-714 Standard Uptake Value ratio (SUVr) in cerebellum
Cytokine and chemokine levels in plasma | 6 months after the last injection
  Luminex magnetic beads technology
PBMC profile | 6 months after the last injection
  High-dimensional characterization of immune reprogramming during the treatment by single-cell RNA-sequencing of PBMC.
Transcriptomics and regulatory epigenomics of circulating monocytes and lymphocytes 1. | 6 months after the last injection
  H3K27ac
Transcriptomics and regulatory epigenomics of circulating monocytes and lymphocytes 2. | 6 months after the last injection
  H3K4me3
Transcriptomics and regulatory epigenomics of circulating monocytes and lymphocytes 3. | 6 months after the last injection
  ChIP-seq
Transcriptomics and regulatory epigenomics of circulating monocytes and lymphocytes 4. | 6 months after the last injection
  ATAC-seq
Genome-wide single-nucleotide polymorphism (SNP) genotype. | After 1 injection
  DNA sample

OTHER OUTCOMES:
Analyze the pharmacokinetics and pharmacodynamics of CSM WJ-UC in humans 1 | After 3rd injection 48 hours later
  NGS approach,
Analyze the pharmacokinetics and pharmacodynamics of CSM WJ-UC in humans 2 | After 3rd injection 48 hours later
  digital droplet (dd)-PCR approach,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 1 | After 3rd injection 48 hours later
  populations of immune effector cells, such as Tregs,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration.2 | After 3rd injection 48 hours later
  populations of immune effector cells, such as Teff,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration.3 | After 3rd injection 48 hours later
  populations of immune effector cells, such as NK cells,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 4 | After 3rd injection 48 hours later
  populations of immune effector cells, such as NKT,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 5 | After 3rd injection 48 hours later
  populations of immune effector cells, such as MAIT,
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 6 | After 3rd injection 48 hours later
  populations of immune effector cells, such as DC
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 7 | After 3rd injection 48 hours later
  populations of immune effector cells, such as monocytes
Deep phenotyping of the main immune effector cell populations humans, to identify the phenotypes involved in immunomodulation and alloimmunization induced by MSC administration. 8 | After 3rd injection 48 hours later
  populations of immune effector cells, such as B cells.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DEGOS, Principal Investigator — APHP
Locations (3):
- France (3):
  - Hôpital National d'Instruction des Armées Percy, Clamart
  - Beaujon Hospital, Clichy
  - Hôpital de la Pitié Salpêtrière - AP-HP, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sigaut S, Tardivon C, Jacquens A, Bottlaender M, Gervais P, Habert MO, Monsel A, Roquilly A, Boutonnet M, Galanaud D, Cras A, Boucher-Pillet H, Florence AM, Cavalier I, Menasche P, Degos V, Couffignal C. Effects of intravascular administration of mesenchymal stromal cells derived from Wharton's Jelly of the umbilical cord on systemic immunomodulation and neuroinflammation after traumatic brain injury (TRAUMACELL): study protocol for a multicentre randomised controlled trial. BMJ Open. 2024 Dec 31;14(12):e091441. doi: 10.1136/bmjopen-2024-091441. PMID 39740941